CLINICAL TRIAL: NCT01565551
Title: Transforming Research and Clinical Knowledge in Traumatic Brain Injury Pilot
Brief Title: Transforming Research and Clinical Knowledge in TBI Pilot
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: RC2NS069409 (NIH); RC2NS069409 (NIH)
Record Dates: First submitted 2012-03-24; First posted 2012-03-28 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Common Data Elements; Prognostic Models; Neuroimaging; Biomarkers; Genetic Variants; Concussion; Psychological Health
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Psychological Well-Being | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for genetic analysis. Plasma for proteomic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early-Presenting TBI: Acute Sites: This cohort of patients are studied after acute presentation within 24 hours of TBI to one of the three TRACK-TBI acute Level I Trauma Centers (SFGH, UPMC, UMCB).
  Interventions: Other: N/A (Observational Study)
- Late-Presenting TBI: Rehabilitation Center: This cohort of patients are studied after presentation to the TRACK-TBI rehabilitation site (MSMC).
  Interventions: Other: N/A (Observational Study)

INTERVENTIONS:
Other: N/A (Observational Study) — No Interventions: Observational Study

SUMMARY:
The global aim of this proposal is to test and refine Common Data Elements (CDEs), neuroimaging standards, and best practices for genetics and proteomics in Traumatic Brain Injury (TBI) studies. Testing and validating of TBI-CDEs will be performed in a multi-center prospective observational study with 3 TBI Centers (San Francisco General Hospital (SFGH), University of Pittsburgh Medical Center (UPMC), University Medical Center Brackenridge (UMCB)) and a TBI Rehabilitation Center (Mount Sinai Rehabilitation Center (MSMC)). The investigators will create and expand existing data repositories for patient demographics, neuroimaging, plasma biomarkers, genetics, and multivariate outcomes thereby providing researchers and clinicians with the infrastructure to establish multidisciplinary, multicenter research networks and improve clinical research in the TBI field.

DETAILED DESCRIPTION:
The Investigators aim for a 10-month data collection period for TBI patients across the spectrum from concussion to coma with a limited 3-month follow up and extensive 6-, 12-, and 24-month follow ups. Patient enrollment will occur in three high-volume TBI Centers (SFGH, UPMC, UMCB) and a TBI Rehabilitation Center (MSMC). These Centers have a long track record of multi-center TBI research experience as well as existing infrastructure for rapid start-up and sustained enrollment. All patients admitted acutely with a history of external force injury to the head with a head CT performed in the emergency department are eligible for enrollment. Head CTs are performed according to the American College of Emergency Physicians (ACEP) and the Centers for Disease Control and Prevention (CDC) Guidelines for neuroimaging and decision making in TBI. These Guidelines are already in place at the participating Centers and are used to determine which patients will receive a non-contrast head CT scan as part of their initial evaluation. Patients will not be excluded based on age, race, gender, ethnicity, substance abuse, or prior psychiatric history to provide a population-based sample of of TBI subjects across the injury spectrum from concussion to coma.

Study Components (Ref: NIH-NINDS TBI Common Data Elements):

1. Clinical Care and Demographic Data Collection. Variables include: date and time of injury, mechanism of injury, acute laboratory values and vital signs, neurological evaluations, surgical interventions, hospital course, morbidity and mortality during acute care.
2. Blood Draw for Proteomic and Genetic Marker Analyses. Blood samples will be drawn within 24 hours of injury. Plasma will be spun and separated from whole blood. Both plasma and whole blood samples will be banked centrally under -80 degrees Celsius at the University of California, San Francisco (UCSF) DNA Bank.
3. 3-Tesla (3T) Magnetic Resonance Imaging. A 3T Research MRI will be completed on a subset of patients able to return 1-2 weeks post-injury.
4. 3-Month Follow Up. The Glasgow Outcome Scale - Extended (GOS-E) and neurological symptoms inventory will be administered to patients over the phone 3 months post-injury.
5. 6-, 12-, and 24-Month Neurocognitive Assessment. Standardized measures from all designated CORE domains for outcome after TBI by TBI-CDEs, which include: global recovery, functional outcome, psychological impairment, post-traumatic stress disorder (PTSD), and quality of life, will be administered to the participant.

The investigators anticipate that this project has the potential to substantially advance and revolutionize clinical research in TBI. Repositories for neuroimaging, proteomic, and genetic biomarkers will facilitate the evolving field of these emerging technologies in TBI.

Recent Publications:

Yue JK, Vassar MJ, Lingsma H, Cooper SR, Yuh EL, Mukherjee P, Puccio AM, Gordon W, Okonkwo DO, Valadka A, Schnyer DM, Maas A, Manley GT; TRACK-TBI Investigators. Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) Pilot: Multicenter Implementation of the Common Data Elements for Traumatic Brain Injury. J Neurotrauma. 2013 Nov 15;30(22):1831-44.

Dams-O'Connor K, Spielman L, Singh A, Gordon WA, Lingsma HF, Maas AI, Manley GT, Mukherjee P, Okonkwo DO, Puccio AM, Schnyer DM, Valadka AB, Yue JK, Yuh EL; TRACK-TBI Investigators. The Impact of Prior Traumatic Brain Injury on Health and Functioning: a TRACK-TBI Study. J Neurotrauma. 2013 Dec 15;30(24):2014-20.

McMahon PJ, Hricik AJ, Yue JK, Puccio AM, Inoue T, Lingsma H, Beers SR, Gordon W, Valadka, A, Manley GT, Okonkwo DO; TRACK-TBI Investigators. Symptomatology and Functional Outcome in Mild Traumatic Brain Injury: Results from the Prospective TRACK-TBI Study. J Neurotrauma. 2013 Oct 31. [Epub ahead of print]

Diaz-Arrastia R, Wang KK, Papa L, Sorani MD, Yue JK, Puccio AM, McMahon PJ, Inoue T, Yuh EL, Lingsma H, Maas A, Valadka A, Okonkwo DO, Manley GT; TRACK-TBI Investigators. Acute Biomarkers of Traumatic Brain Injury: Relationship Between Plasma Levels of Ubiquitin C-Terminal Hydrolase-L1 (UCH-L1) and Glial Fibrillary Acidic Protein (GFAP). J Neurotrauma. 2013 Oct 9. [Epub ahead of print]

Okonkwo DO, Yue JK, Puccio AM, Panczykowski D, Inoue T, McMahon PJ, Sorani MD, Yuh EL, Lingsma H, Maas A, Valadka A, Manley GT; TRACK-TBI Investigators. GFAP-BDP as an Acute Diagnostic Marker of Traumatic Brain Injury: Results from the Prospective TRACK-TBI Study. J Neurotrauma. 2013 Sep 1;30(17):1490-7.

Yuh EL, Mukherjee P, Lingsma HF, Yue JK, Ferguson AR, Gordon WA, Valadka AB, Schnyer DM, Okonkwo DO, Maas AI, Manley GT; TRACK-TBI Investigators. Magnetic Resonance Imaging Improves 3-Month Outcome Prediction in Mild Traumatic Brain Injury. Ann Neurol. 2013 Feb;73(2):224-35.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to Emergency Department < 24 hours post-injury
* Head CT scan for Traumatic Brain Injury (TBI) as part of regular care.
* English Speaking

Exclusion Criteria:

* Presentation to Emergency Department > 24 hours post-injury
* Custody or Incarceration
* 5150 Psychiatric Hold

Component-Specific Exclusion Criteria:

MRI: Pregnant or may be pregnant; younger than 8 years old; those who have cardiac pacemakers, neural pacemakers, surgical clips in the brain or blood vessels, surgically implanted metal plates, screws or pins, cochlear implants, intrauterine devices (IUDs), or metal objects in their body, especially in the eye. Persons with a history of claustrophobia are excluded from this procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a population-based TBI study. All patients presenting to the acute sites with traumatic brain injury and receive a head CT scan as part of standard care within 24 hours of injury date and time are initially eligible. As most six-month Common Date Elements (CDE) outcome measures are normed and validated only in English, study participants must be English-speaking. There are no other restrictions to eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey T Manley, MD, PhD, Principal Investigator — University of California, San Francisco (San Francisco, CA); David O Okonkwo, MD, PhD, Principal Investigator — University of Pittsburgh; Alex B Valadka, MD, Principal Investigator — University Medical Center, Brackenridge (Austin, TX); Wayne A Gordon, PhD, Principal Investigator — Mount Sinai Rehabilitation Center (New York, NY)
Locations (4):
- United States (4):
  - San Francisco General Hospital (SFGH), San Francisco, California
  - Mount Sinai Rehabilitation Center, New York, New York
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - University Medical Center, Brackenridge, Austin, Texas

REFERENCES:
- [Background] Finkelstein E, Corso P, Miller T. The Incidence and Economic Burden of Injuries in the United States. New York, NY: Oxford University Press; 2006.
- [Background] Foulkes AM, Eisenberg MH, Jane AJ. The Traumatic Coma Data Bank; design, methods and baseline characteristics. J. Neuroch. 75, S1-S15, 1991
- [Background] Jagoda AS, Bazarian JJ, Bruns JJ Jr, Cantrill SV, Gean AD, Howard PK, Ghajar J, Riggio S, Wright DW, Wears RL, Bakshy A, Burgess P, Wald MM, Whitson RR. Clinical policy: neuroimaging and decisionmaking in adult mild traumatic brain injury in the acute setting. J Emerg Nurs. 2009 Apr;35(2):e5-40. doi: 10.1016/j.jen.2008.12.010. PMID 19285163
- [Background] Maas AI, Stocchetti N, Bullock R. Moderate and severe traumatic brain injury in adults. Lancet Neurol. 2008 Aug;7(8):728-41. doi: 10.1016/S1474-4422(08)70164-9. PMID 18635021
- [Background] Marmarou A, Lu J, Butcher I, McHugh GS, Mushkudiani NA, Murray GD, Steyerberg EW, Maas AI. IMPACT database of traumatic brain injury: design and description. J Neurotrauma. 2007 Feb;24(2):239-50. doi: 10.1089/neu.2006.0036. PMID 17375988
- [Background] Marshall LF, Marshall SB, Klauber MR, Van Berkum Clark M, Eisenberg H, Jane JA, Luerssen TG, Marmarou A, Foulkes MA. The diagnosis of head injury requires a classification based on computed axial tomography. J Neurotrauma. 1992 Mar;9 Suppl 1:S287-92. PMID 1588618
- [Background] MRC CRASH Trial Collaborators; Perel P, Arango M, Clayton T, Edwards P, Komolafe E, Poccock S, Roberts I, Shakur H, Steyerberg E, Yutthakasemsunt S. Predicting outcome after traumatic brain injury: practical prognostic models based on large cohort of international patients. BMJ. 2008 Feb 23;336(7641):425-9. doi: 10.1136/bmj.39461.643438.25. Epub 2008 Feb 12. PMID 18270239
- [Background] Murray GD, Teasdale GM, Braakman R, Cohadon F, Dearden M, Iannotti F, Karimi A, Lapierre F, Maas A, Ohman J, Persson L, Servadei F, Stocchetti N, Trojanowski T, Unterberg A. The European Brain Injury Consortium survey of head injuries. Acta Neurochir (Wien). 1999;141(3):223-36. doi: 10.1007/s007010050292. PMID 10214478
- [Background] Ng J, Wahl M, Tong L, Lee H, Veeraraghavan S, Xu D, Zhao S, Kornak J, Meeker M, Ghajar J, Manley GT, Mukherjee P. 3T Diffusion Tensor Imaging of Mild Traumatic Brain Injury: A Prospective Longitudinal Study. Proc ISMRM 2009; 641.
- [Background] Niogi SN, Mukherjee P, Ghajar J, Johnson CE, Kolster R, Lee H, Suh M, Zimmerman RD, Manley GT, McCandliss BD. Structural dissociation of attentional control and memory in adults with and without mild traumatic brain injury. Brain. 2008 Dec;131(Pt 12):3209-21. doi: 10.1093/brain/awn247. Epub 2008 Oct 24. PMID 18952679
- [Background] Saatman KE, Duhaime AC, Bullock R, Maas AI, Valadka A, Manley GT; Workshop Scientific Team and Advisory Panel Members. Classification of traumatic brain injury for targeted therapies. J Neurotrauma. 2008 Jul;25(7):719-38. doi: 10.1089/neu.2008.0586. PMID 18627252
- [Background] Steyerberg EW, Mushkudiani N, Perel P, Butcher I, Lu J, McHugh GS, Murray GD, Marmarou A, Roberts I, Habbema JD, Maas AI. Predicting outcome after traumatic brain injury: development and international validation of prognostic scores based on admission characteristics. PLoS Med. 2008 Aug 5;5(8):e165; discussion e165. doi: 10.1371/journal.pmed.0050165. PMID 18684008
- [Background] Rusnak M, Janciak I, Majdan M, Wilbacher I, Mauritz W; Australian Severe TBI Study Investigators. Severe traumatic brain injury in Austria VI: effects of guideline-based management. Wien Klin Wochenschr. 2007 Feb;119(1-2):64-71. doi: 10.1007/s00508-006-0765-0. PMID 17318752
- [Background] Wakana S, Caprihan A, Panzenboeck MM, Fallon JH, Perry M, Gollub RL, Hua K, Zhang J, Jiang H, Dubey P, Blitz A, van Zijl P, Mori S. Reproducibility of quantitative tractography methods applied to cerebral white matter. Neuroimage. 2007 Jul 1;36(3):630-44. doi: 10.1016/j.neuroimage.2007.02.049. Epub 2007 Mar 20. PMID 17481925
- [Background] Yuh EL, Gean AD, Manley GT, Callen AL, Wintermark M. Computer-aided assessment of head computed tomography (CT) studies in patients with suspected traumatic brain injury. J Neurotrauma. 2008 Oct;25(10):1163-72. doi: 10.1089/neu.2008.0590. PMID 18986221
- [Derived] Yue JK, Kobeissy FH, Jain S, Sun X, Phelps RRL, Korley FK, Gardner RC, Ferguson AR, Huie JR, Schneider ALC, Yang Z, Xu H, Lynch CE, Deng H, Rabinowitz M, Vassar MJ, Taylor SR, Mukherjee P, Yuh EL, Markowitz AJ, Puccio AM, Okonkwo DO, Diaz-Arrastia R, Manley GT, Wang KKW. Neuroinflammatory Biomarkers for Traumatic Brain Injury Diagnosis and Prognosis: A TRACK-TBI Pilot Study. Neurotrauma Rep. 2023 Mar 24;4(1):171-183. doi: 10.1089/neur.2022.0060. eCollection 2023. PMID 36974122
- [Derived] Yue JK, Cnossen MC, Winkler EA, Deng H, Phelps RRL, Coss NA, Sharma S, Robinson CK, Suen CG, Vassar MJ, Schnyer DM, Puccio AM, Gardner RC, Yuh EL, Mukherjee P, Valadka AB, Okonkwo DO, Lingsma HF, Manley GT; TRACK-TBI Investigators. Pre-injury Comorbidities Are Associated With Functional Impairment and Post-concussive Symptoms at 3- and 6-Months After Mild Traumatic Brain Injury: A TRACK-TBI Study. Front Neurol. 2019 Apr 9;10:343. doi: 10.3389/fneur.2019.00343. eCollection 2019. PMID 31024436
- [Derived] Ranson J, Magnus BE, Temkin N, Dikmen S, Giacino JT, Okonkwo DO, Valadka AB, Manley GT, Nelson LD; TRACK-TBI Investigators. Diagnosing the GOSE: Structural and Psychometric Properties Using Item Response Theory, a TRACK-TBI Pilot Study. J Neurotrauma. 2019 Sep 1;36(17):2493-2505. doi: 10.1089/neu.2018.5998. Epub 2019 May 23. PMID 30907261
- [Derived] Yue JK, Winkler EA, Sharma S, Vassar MJ, Ratcliff JJ, Korley FK, Seabury SA, Ferguson AR, Lingsma HF, Deng H, Meeuws S, Adeoye OM, Rick JW, Robinson CK, Duarte SM, Yuh EL, Mukherjee P, Dikmen SS, McAllister TW, Diaz-Arrastia R, Valadka AB, Gordon WA, Okonkwo DO, Manley GT; the TRACK-TBI Investigators. Temporal profile of care following mild traumatic brain injury: predictors of hospital admission, follow-up referral and six-month outcome. Brain Inj. 2017;31(13-14):1820-1829. doi: 10.1080/02699052.2017.1351000. PMID 29166203
- [Derived] Nelson LD, Ranson J, Ferguson AR, Giacino J, Okonkwo DO, Valadka AB, Manley GT, McCrea MA. Validating Multi-Dimensional Outcome Assessment Using the Traumatic Brain Injury Common Data Elements: An Analysis of the TRACK-TBI Pilot Study Sample. J Neurotrauma. 2017 Nov 15;34(22):3158-3172. doi: 10.1089/neu.2017.5139. Epub 2017 Aug 17. PMID 28595478
- [Derived] Nielson JL, Cooper SR, Yue JK, Sorani MD, Inoue T, Yuh EL, Mukherjee P, Petrossian TC, Paquette J, Lum PY, Carlsson GE, Vassar MJ, Lingsma HF, Gordon WA, Valadka AB, Okonkwo DO, Manley GT, Ferguson AR; TRACK-TBI Investigators. Uncovering precision phenotype-biomarker associations in traumatic brain injury using topological data analysis. PLoS One. 2017 Mar 3;12(3):e0169490. doi: 10.1371/journal.pone.0169490. eCollection 2017. PMID 28257413
- [Derived] Yue JK, Winkler EA, Rick JW, Burke JF, McAllister TW, Oh SS, Burchard EG, Hu D, Rosand J, Temkin NR, Korley FK, Sorani MD, Ferguson AR, Lingsma HF, Sharma S, Robinson CK, Yuh EL, Tarapore PE, Wang KK, Puccio AM, Mukherjee P, Diaz-Arrastia R, Gordon WA, Valadka AB, Okonkwo DO, Manley GT; TRACK-TBI Investigators. DRD2 C957T polymorphism is associated with improved 6-month verbal learning following traumatic brain injury. Neurogenetics. 2017 Jan;18(1):29-38. doi: 10.1007/s10048-016-0500-6. Epub 2016 Nov 8. PMID 27826691
- [Derived] Winkler EA, Yue JK, McAllister TW, Temkin NR, Oh SS, Burchard EG, Hu D, Ferguson AR, Lingsma HF, Burke JF, Sorani MD, Rosand J, Yuh EL, Barber J, Tarapore PE, Gardner RC, Sharma S, Satris GG, Eng C, Puccio AM, Wang KK, Mukherjee P, Valadka AB, Okonkwo DO, Diaz-Arrastia R, Manley GT; TRACK-TBI Investigators. COMT Val 158 Met polymorphism is associated with nonverbal cognition following mild traumatic brain injury. Neurogenetics. 2016 Jan;17(1):31-41. doi: 10.1007/s10048-015-0467-8. Epub 2015 Nov 17. PMID 26576546
- [Derived] McMahon PJ, Panczykowski DM, Yue JK, Puccio AM, Inoue T, Sorani MD, Lingsma HF, Maas AI, Valadka AB, Yuh EL, Mukherjee P, Manley GT, Okonkwo DO; TRACK-TBI Investigators. Measurement of the glial fibrillary acidic protein and its breakdown products GFAP-BDP biomarker for the detection of traumatic brain injury compared to computed tomography and magnetic resonance imaging. J Neurotrauma. 2015 Apr 15;32(8):527-33. doi: 10.1089/neu.2014.3635. Epub 2015 Jan 26. PMID 25264814
- [Derived] Lingsma HF, Yue JK, Maas AI, Steyerberg EW, Manley GT; TRACK-TBI Investigators. Outcome prediction after mild and complicated mild traumatic brain injury: external validation of existing models and identification of new predictors using the TRACK-TBI pilot study. J Neurotrauma. 2015 Jan 15;32(2):83-94. doi: 10.1089/neu.2014.3384. Epub 2014 Nov 25. PMID 25025611
- [Derived] Ratcliff JJ, Adeoye O, Lindsell CJ, Hart KW, Pancioli A, McMullan JT, Yue JK, Nishijima DK, Gordon WA, Valadka AB, Okonkwo DO, Lingsma HF, Maas AI, Manley GT; TRACK-TBI investigators. ED disposition of the Glasgow Coma Scale 13 to 15 traumatic brain injury patient: analysis of the Transforming Research and Clinical Knowledge in TBI study. Am J Emerg Med. 2014 Aug;32(8):844-50. doi: 10.1016/j.ajem.2014.04.003. Epub 2014 Apr 13. PMID 24857248
- [Derived] McMahon P, Hricik A, Yue JK, Puccio AM, Inoue T, Lingsma HF, Beers SR, Gordon WA, Valadka AB, Manley GT, Okonkwo DO; TRACK-TBI Investigators. Symptomatology and functional outcome in mild traumatic brain injury: results from the prospective TRACK-TBI study. J Neurotrauma. 2014 Jan 1;31(1):26-33. doi: 10.1089/neu.2013.2984. Epub 2013 Oct 31. PMID 23952719
- [Derived] Dams-O'Connor K, Spielman L, Singh A, Gordon WA, Lingsma HF, Maas AI, Manley GT, Mukherjee P, Okonkwo DO, Puccio AM, Schnyer DM, Valadka AB, Yue JK, Yuh EL; TRACK-TBI Investigators. The impact of previous traumatic brain injury on health and functioning: a TRACK-TBI study. J Neurotrauma. 2013 Dec 15;30(24):2014-20. doi: 10.1089/neu.2013.3049. Epub 2013 Oct 23. PMID 23924069
- [Derived] Diaz-Arrastia R, Wang KK, Papa L, Sorani MD, Yue JK, Puccio AM, McMahon PJ, Inoue T, Yuh EL, Lingsma HF, Maas AI, Valadka AB, Okonkwo DO, Manley GT; TRACK-TBI Investigators. Acute biomarkers of traumatic brain injury: relationship between plasma levels of ubiquitin C-terminal hydrolase-L1 and glial fibrillary acidic protein. J Neurotrauma. 2014 Jan 1;31(1):19-25. doi: 10.1089/neu.2013.3040. Epub 2013 Oct 9. PMID 23865516
- [Derived] Yue JK, Vassar MJ, Lingsma HF, Cooper SR, Okonkwo DO, Valadka AB, Gordon WA, Maas AI, Mukherjee P, Yuh EL, Puccio AM, Schnyer DM, Manley GT; TRACK-TBI Investigators. Transforming research and clinical knowledge in traumatic brain injury pilot: multicenter implementation of the common data elements for traumatic brain injury. J Neurotrauma. 2013 Nov 15;30(22):1831-44. doi: 10.1089/neu.2013.2970. Epub 2013 Sep 24. PMID 23815563
- [Derived] Okonkwo DO, Yue JK, Puccio AM, Panczykowski DM, Inoue T, McMahon PJ, Sorani MD, Yuh EL, Lingsma HF, Maas AI, Valadka AB, Manley GT; Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) Investigators. GFAP-BDP as an acute diagnostic marker in traumatic brain injury: results from the prospective transforming research and clinical knowledge in traumatic brain injury study. J Neurotrauma. 2013 Sep 1;30(17):1490-7. doi: 10.1089/neu.2013.2883. Epub 2013 Aug 1. PMID 23489259

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early-Presenting TBI: Acute Sites | Late-Presenting TBI: Rehabilitation Center
Started | 586 | 51
Clinical/Demographics | 586 | 51
Biospecimens/Biomarkers | 479 | 22
Neuroimaging | 233 | 25
6-Month Outcomes | 412 | 30
Completed | 586 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-Presenting TBI: Acute Sites | Late-Presenting TBI: Rehabilitation Center | Total
Number analyzed (Participants) | 586 | 51 | 637
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.3 (18.5) | 49.9 (20.4) | 43.9 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 14 | 181
  Male | 419 | 37 | 456
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 22 | 2 | 24
  Native Hawaiian or Other Pacific Islander | 17 | 0 | 17
  Black or African American | 46 | 9 | 55
  White | 471 | 39 | 510
  More than one race | 21 | 0 | 21
  Unknown or Not Reported | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 84 | 5 | 89
  Not Hispanic or Latino | 495 | 33 | 528
  Unknown or Not Reported | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Glasgow Outcome Scale Extended (GOSE)
Description: The GOSE provides and overall measure of disability based on information on cognition, independence, employability, and social/community participation collected via structured interview. Individuals are described by one of the eight outcome categories: Dead (1); Vegetative State (2); Lower Severe Disability (3); Upper Severe Disability (4); Lower Moderate Disability (5); Upper Moderate Disability (6); Lower Good Recovery (7) and Upper Good Recovery (8). Good Recovery is defined as a score of 7-8, Moderate Disability is defined by a score of 5-6 and Severe Disability is defined by a score of 3-4.
Time Frame: 6 Months Post-Injury
Measure: Median (Inter-Quartile Range); unit: Glasgow Outcome Scale Extended (GOSE)
Arm/Group | Early-Presenting TBI: Acute Sites | Late-Presenting TBI: Rehabilitation Center
Number analyzed (Participants) | 414 | 28
Glasgow Outcome Scale Extended (GOSE) | 7 [5 to 8] | 5 [4 to 7]

ADVERSE EVENTS:
Time Frame: 6 Months Post-Injury
Arm/Group | Early-Presenting TBI: Acute Sites | Late-Presenting TBI: Rehabilitation Center
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Enrolling patients representative of the TBI population created challenges for follow-up (e.g. homelessness, substance abuse); limited access to research MRI scanner; lack of validated outcome measures for non-English-speaking and pediatric patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No